CLINICAL TRIAL: NCT04860453
Title: Genomic Analysis of Families With a History of Discordant Cancers
Status: Recruiting | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: CASE13Z20
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Discordant Cancers
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Affected participants with 5 or more discordant cancers - WES: Affected individuals with a family history of 5 or more discordant cancers in unilateral descent with a 3-generation pedigree will receive SOC CLIA/CAP multicancer panel (DNA collected via blood draw or punch biopsy) to examine monogenic variant diagnostic yield. Eligible participants (families with no mutations and at least 2 affected and 1 non-affected family members) may move forward with WES.
  Any identified monogenic variants of interest will be sent to an industry partner with CLIA/CAP certification for validation. A 6-month follow-up visit will take place during which variants will be discussed and participants who underwent gHFI variant counting (those who were not considered a gene candidate) will have results explained. Appropriate genetic counselling, recurrence risk, and additional clinical referrals will be made as necessary
  Interventions: Genetic: WES via Illumina NextSeq 550 sequencing system; Diagnostic Test: Blood Draw; Diagnostic Test: Skin biopsy; Diagnostic Test: Saliva Sample
- SOC genetic counseling (routine clinical care): Affected individuals (cancer) with a family history suggestive of a known hereditary syndrome or meeting NCCN criteria for germline testing will receive SOC CLIA/CAP multicancer panel in order to examine monogenic variant diagnostic yield (retrospective data)
  This arm would also include prospective participants from the "5 or more discordant cancers" group who DID have a variant identified and therefore did not move on to WES.
  Interventions: Diagnostic Test: Blood Draw; Diagnostic Test: Skin biopsy; Diagnostic Test: Saliva Sample

INTERVENTIONS:
Genetic: WES via Illumina NextSeq 550 sequencing system — Sequencing will be performed on an Illumina sequencing system
  Groups: Affected participants with 5 or more discordant cancers - WES
Diagnostic Test: Blood Draw — Blood draw will be via any University Hospitals Laboratory site and sent at room temperature via courier to the Center for Human Genetics (CHG) Laboratory
Diagnostic Test: Skin biopsy — Skin samples obtained via 3mm punch biopsy will be suspended in cell culture media prepared per CHG routine and sent via courier to the Center for Human Genetics Laboratory
Diagnostic Test: Saliva Sample — Participant will provide a saliva sample which be shipped to University Hospitals Laborator site at room temperature

SUMMARY:
The purpose of this study is to identify novel gene mutations which have contributed to significant personal and family history of cancer. Adults with and without cancer will be accrued to the study. Participants qualify to take part in this research study because someone in their family has been diagnosed with or because they themselves have a cancer diagnosis.

Participants' DNA and other clinical information will be obtained from a blood sample in order to study the genetic basis of cancer and related complications. All portions in the DNA that code for proteins (i.e., the exome) will be studied. Participant DNA sample and information about family structure and family medical history and ethnic origin may also be collected to better understand this information. Clinical information will be stored and biological samples, including DNA, will be kept for up to three (3) years after collection for future. Ultimately, once identified, the role of the specific genetics changes in the development of inherited cancer(s) will be characterized.

DETAILED DESCRIPTION:
Data for this study will be obtained via both retrospectively and prospectively. Affected individuals (who have cancer) with a family history suggestive of a known hereditary syndrome or meeting National Comprehensive Cancer Network (NCCN) criteria will be accrued from routine clinical care to form a "real world" baseline of diagnostic yield using a multicancer panel. These participants will not be additionally consented for WES as part the clinical study.

Other affected individuals identified as having five or more relatives with discordant cancers will receive standard of care (SOC) multicancer panel. Families without any mutations identified (with at least a minimum of 2 members with cancer, 1 without) will be considered for additional sequencing as part of this study's primary objective of describing novel inherited cancer syndromes.

If the individual being evaluated in cancer genetics clinic (i.e. index patient) consents and their family members express interest in the study, they will move on to study visit 1. During this visit, pedigree information and medical histories will be explained, consent verified, and individual genetic counselling provided. Individuals will decide whether or not to be notified that incidental findings exist in their genomes.

Lab requisition will be done to facilitate blood draws and DNA extraction/storage and WES analysis will be completed. Any identified monogenic variants of interest will be sent to an industry partner with Clinical Laboratory Improvement Amendments (CLIA)/College of American Pathologists (CAP) certification for validation.

Study visit 2 to be completed within the next 6 months, at which any identified monogenetic variants of interest will be discussed with the participant. Those undergoing Germline High Functional Impact (gHFI) variant counting will be notified if they have more or less than the general population. Appropriate genetic counselling, recurrence risk, and additional clinical referrals will be made as necessary. Participants will be notified with a binary yes/no of any American College of Medical Genetics incidental findings and a routine clinical genetics follow-up appointment will be made

The primary objective of the study is to identify novel gene variants associated with generalized cancer susceptibility that is manifesting as a personal history of multiple primary tumors or a family history of discordant cancers. This will be done through exploratory, research grade (ie NOT CLIA/CAP certified) whole exome sequencing (WES) studies provided to patients/families with family histories of discordant cancers as an adjunct to SOC clinical genetics evaluation in order to clinically describe novel syndromic manifestations of cancer susceptibility. Suspected germline variants supporting a generalized cancer susceptibility will be further validated in a CLIA/CAP certified laboratory prior to being reported out to the patient's medical chart

ELIGIBILITY:
Inclusion Criteria:

* Affected patient with a family history suggestive of a known hereditary syndrome or meeting NCCN criteria for germline testing and consent to a multicancer panel

  --This cohort is meant as a real world control group receiving routine standard of care and is not eligible for WES.
* Affected patient with a family history of 5 or more discordant cancers in unilateral descent within a 3-generation pedigree.

  * Unaffected family members within such kindreds will be eligible for WES as long as a minimum of 2 affected and 1 unaffected family members consent to WES as trial participants.

Exclusion Criteria:

* Unable to safely provide a blood sample for genetic testing
* Unable to receive or decline to receive genetic counselling through the telephone, video conference, or in person
* Families known to segregate a previously identified high penetrance cancer susceptibility gene identified through routine medical genetics evaluation are not eligible WES
* Family is not amenable to routine medical genetics SOC genetics evaluation.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Family history suggestive of a known hereditary cancer syndrome
  2. 5 or more relatives with discordant cancer diagnoses
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-11-17 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a family history of 5 or more discordant cancers that have monogenic germline variants identifiable with WES sequencing | At baseline for an average of 1.5 hours
  Number of participants with a family history of 5 or more discordant cancers that have monogenic germline variants identifiable with WES sequencing
  The diagnostic yield of monogenic germline variants will be calculated as the discovery rate for a monogenic pathogenic variant within each category (ie 10 pathogenic variants / 30 families = 33% yield rate).
  A 2-way ANOVA will be performed, with the null hypothesis being that "family history supportive of a known syndrome versus discordant cancers does not significantly affect diagnostic yield"
Number of gHFI variants | At baseline for an average of 1.5 hours
  Number of gHFI variants in participants with a family history of 5 or more discordant and no identified monogenic pathogenic germline variants on WES compared to population averages
  Number of gHFI variants in family members within such kindreds and no cancer diagnoses will compared to those with cancer diagnoses
Diagnostic yield for monogenic germline variants in two arms | At baseline for an average of 1.5 hours
  Diagnostic yield for monogenic germline variants in arm I (routine real-world clinical practice) vs arm II (5 or more relatives with discordant cancer diagnoses) using multicancer panels
  The diagnostic yield of monogenic germline variants will be calculated as the discovery rate for a monogenic pathogenic variant within each category (ie 10 pathogenic variants / 30 families = 33% yield rate).
  A 2-way ANOVA will be performed, with the null hypothesis being that "family history supportive of a known syndrome versus discordant cancers does not significantly affect diagnostic yield"

CONTACTS AND LOCATIONS:
Overall Officials: Anna Mitchell, MD PhD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Due to privacy concerns of family history and genetic information of data collected, individual participant data (IPD) will not be shared